CLINICAL TRIAL: NCT00063648
Title: Detection and Cytotoxic T Lymphocyte Therapy of Post-Transplant Lymphoproliferative Disorder After Liver Transplant
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PTLD (completed)
Record Dates: First submitted 2003-07-01; First posted 2003-07-03 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2010-01

CONDITIONS: Liver Disease; Lymphoproliferative Disorders
Keywords: PTLD; CTL Therapy; Post-transplant lymphoproliferative disorder
MeSH Terms: conditions — Liver Diseases; Lymphoproliferative Disorders

INTERVENTIONS:
Biological: EBV-specific autologous CTL

SUMMARY:
Despite advances in medical and gene therapy, orthotopic liver transplantation remains the only definitive therapeutic option for children with end-stage liver disease. Recent advances in pre-, intra-, and early post-transplant care have resulted in a dramatic improvement in survival of the pediatric liver transplant patient. The broad long-range goal of our research program is directed at enhancing the patient's long-term survival. Our primary focus relates to obligate life-long immunosuppression, with its inherent complications including severe infection and development of cancer. These two complications come together in a single disease, Epstein-Barr Virus (EBV)- associated post-transplant lymphoproliferative disorder (PTLD). EBV, a latent human lymphotrophic herpes virus infects and immortalizes B cells. Primary infection usually occurs via salivary exchange and results in a mild, self-limited illness followed by life-long EBV-specific T cell controlled EBV latency. T cell-based immunosuppression prevents allograft rejection, however, it also suppresses cytotoxic T lymphocyte (CTL) function, generating an environment in which EBV-infected cells can proliferate. Patients receiving life-long T cell-based immunosuppression have an increased risk of developing PTLD due to their inability to produce normal immunoregulatory responses. This disease is particularly devastating to the pediatric patient as its incidence is at least 4-fold greater than in the adult liver transplant patient population. In fact, PTLD is the number one cause of death following pediatric liver transplantation. At this time, there is no definitive method of prospectively detecting, diagnosing, or treating PTLD, and current treatment protocols place the liver allograft and patient at risk. Therefore, a diagnostic tool that is both sensitive and specific, and a treatment strategy with low toxicity are greatly needed to decrease the morbidity and mortality suffered by the pediatric liver transplant patient with PTLD. Our proposed studies will support our hypothesis that the combination of a persistently elevated EBV load in the setting of a diminished immune response to EBV will be an early risk indicator associated with PTLD development, and that pre-emptive treatment utilizing autologous adoptive EBV-specific CTL immunotherapy will provide a low toxicity treatment option.

ELIGIBILITY:
Pediatric patients s/p orthotopic liver transplantation

Ages: 1 Month to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50
Dates: Start 2002-05; Study Completion 2007-12

CONTACTS AND LOCATIONS:
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States